CLINICAL TRIAL: NCT01242787
Title: A Multinational, Multi-center, Open, Comparative, Paralleled, Roll-over Study to Assess the Safety and Antiviral Activity of LB80380 Tablet Compared to Entecavir 0.5 mg After Additional 48 Weeks of Treatment in Chronic Hepatitis B Patients Who Have Completed LG-BVCL007 Study
Brief Title: Long-term Safety and Efficacy Study of LB80380 in the Treatment-naive Patients of Chronic Hepatitis B
Acronym: LB80380
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BVCL008
Record Dates: First submitted 2010-11-12; First posted 2010-11-17 (Estimated); Last update posted 2012-04-16 (Estimated); Status verified 2012-04

CONDITIONS: Chronic Hepatitis B
Keywords: Chronic hepatitis B; LB80380; treatment-naive; entecavir; Extension
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — ((1-((2-amino-9H-purin-9-yl)methyl)cyclopropyl)oxy)methylphosphonic acid dipivoxyl; entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Entecavir 0.5 mg (Active Comparator): Entecavir 0.5 mg
  Interventions: Drug: Entecavir 0.5 mg
- LB80380 (Experimental): Optimal dose of LB80380 (optimal dose will be chosen early 2011 based on the results of LG-BVCL007 study)
  Interventions: Drug: LB80380

INTERVENTIONS:
Drug: LB80380 — Optimal dose of LB80380, by oral for 48 weeks (optimal dose will be chosen early 2011 based on the results of LG-BVCL007 study)
  Arms: LB80380
Drug: Entecavir 0.5 mg — Entecavir 0.5 mg, by oral for 48 weeks
  Arms: Entecavir 0.5 mg

SUMMARY:
The purpose of the study is to investigate the long-term safety and the antiviral activity of the optimal doses of LB80380 for additional 48 weeks in treatment-naive patients with chronic hepatitis B infection compared to entecavir 0.5 mg.

DETAILED DESCRIPTION:
LB80380, an oral prodrug, is a promising candidate nucleotide analogue with antiviral activity against wild-type hepatitis B virus (HBV). LB80380 is undergoing clinical development by LG Life Sciences for use in the treatment of chronic HBV infection.

This study is an extension study of the Phase IIb (Protocol No. LG-BVCL007), the treatment period of this study is 48-week with 24-week of follow-up period

ELIGIBILITY:
Inclusion Criteria:

* The patients who are able to participate in this expanded study without any interruption after completing 48 weeks treatment of LG-BVCL007 study

Exclusion Criteria:

* Co-infection with hepatitis C or D virus (HCV or HDV) or HIV
* Decompensated liver disease
* ALT > 10 x ULN
* Creatinine clearance (calculated by cockcroft-gault formula) less than 50 ml/min
* Alpha-fetoprotein (AFP) value greater than or equal to 50 ng/mL, and a follow-up ultrasonography performed prior to baseline shows findings indicative of HCC
* Treatment with immunomodulatory agent or corticosteroids within 6 months prior to study entry.
* Pregnancy or breast-feeding
* Patient is currently abusing alcohol or illicit drugs
* Significant systemic illnesses other than liver diseases
* Presence of other causes of liver disease
* Plan for liver transplantation

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2010-08; Primary Completion 2012-09 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients showing HBV DNA mutation | at Week 48
  Safety assessment including adverse events, laboratory abnormalities and DNA mutation

SECONDARY OUTCOMES:
Change of HBV DNA from Baseline of LG-BVCL007 study | at Week 48
  Efficacy assessment including normalization of ALT, HBsAg seroconversion, HBeAg seroconversion

CONTACTS AND LOCATIONS:
Locations (2):
- Queen Mary Hospital, Hong Kong, China
- Severance Hospital of Yonsei University and other 8 sites in Korea, Seoul, South Korea

REFERENCES:
- [Result] Fung J, Lai CL, Yuen MF. LB80380: a promising new drug for the treatment of chronic hepatitis B. Expert Opin Investig Drugs. 2008 Oct;17(10):1581-8. doi: 10.1517/13543784.17.10.1581. PMID 18808318
- [Result] Yuen MF, Lee SH, Kang HM, Kim CR, Kim J, Ngai V, Lai CL. Pharmacokinetics of LB80331 and LB80317 following oral administration of LB80380, a new antiviral agent for chronic hepatitis B (CHB), in healthy adult subjects, CHB patients, and mice. Antimicrob Agents Chemother. 2009 May;53(5):1779-85. doi: 10.1128/AAC.01290-08. Epub 2009 Feb 17. PMID 19223649
- [Result] Yuen MF, Han KH, Um SH, Yoon SK, Kim HR, Kim J, Kim CR, Lai CL. Antiviral activity and safety of LB80380 in hepatitis B e antigen-positive chronic hepatitis B patients with lamivudine-resistant disease. Hepatology. 2010 Mar;51(3):767-76. doi: 10.1002/hep.23462. PMID 20091678
- [Result] Yuen MF, Kim J, Kim CR, Ngai V, Yuen JC, Min C, Kang HM, Shin BS, Yoo SD, Lai CL. A randomized placebo-controlled, dose-finding study of oral LB80380 in HBeAg-positive patients with chronic hepatitis B. Antivir Ther. 2006;11(8):977-83. PMID 17302367